CLINICAL TRIAL: NCT03704272
Title: Supervisory Neglect, Non-Accidental Trauma, Brief Intervention, and Treatment Referral (SunBrite)
Brief Title: Supervisory Neglect, Non-Accidental Trauma, Brief Intervention, and Treatment Referral
Acronym: SunBrite
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was never initiated. No IRB approval obtained, and no participants enrolled.
Sponsor: Phoenix Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-151
Record Dates: First submitted 2018-10-08; First posted 2018-10-12 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: Neglect, Child; Non-Accidental Trauma; Non-Accidental Injury to Child; Head Trauma
MeSH Terms: conditions — Craniocerebral Trauma

STUDY DESIGN:
Intervention Model Description: Control group (Treatment as usual) vs. Treatment group (screening, brief intervention and referral to treatment)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Families in the control group will receive treatment as usual, which includes reporting to child welfare agencies when appropriate.
- Treatment (Experimental): SunBrite
  Interventions: Behavioral: SunBrite

INTERVENTIONS:
Behavioral: SunBrite — SunBrite is a family-empowered injury risk mitigation intervention with 3 core components: screening for the risk of supervisory neglect associated with traumatic injury in very young children; a brief behavioral intervention using motivational interviewing designed to provide feedback to the caregiver on supervisory risk and traumatic injury; and a referral to treatment for ongoing risks such as substance abuse, trauma or mental illness, requiring specific clinical interventions.
  Arms: Treatment

SUMMARY:
The Supervisory Neglect, Non-Accidental Trauma, Brief Intervention, and Treatment Referral (SunBrite) protocol is a family-empowered, risk mitigation strategy that targets families with young children who present to the ED with intracranial trauma. Based on the widely utilized screening, brief intervention, and referral to treatment (SBIRT) protocol, SunBrite has 3 core components: screening, brief motivational interview, and referral for treatment. PCH will: 1) engage community partnerships to support SunBrite development; 2) utilize participatory action research approach for design, implementation, process evaluation, and dissemination of the pilot program; and 3) evaluate intervention implementation and pilot outcomes. Over a 2-year period, this study will encompass a pilot intervention and implementation assessment and a randomized trial to evaluate outcomes. Implementation of SunBrite will yield rigorous scientific evidence for a sustainable, evidenced-based, widely-needed non-accidental (NAT) screening and intervention for families with young children.

DETAILED DESCRIPTION:
SunBrite is a novel, evidence-based intervention for non-accidental trauma (NAT) that has not, as yet, been implemented in any health care setting. Current programs targeting NAT vary widely, and there is insufficient research to conclude that these efforts have reduced re-admission rates(12,13). EDs primarily screen for risk factors associated with child abuse, focusing on their role in reporting and developing forensic evidence for investigations but not on risk reduction. While such efforts as embedding child protection teams in trauma programs are a starting point, much more needs to be done to develop a standard of care and empirically demonstrate efforts that reduce the risk of subsequent injury.

The overlap between non-accidental trauma (NAT) and inadequate caregiver supervision provides an opportunity to identify and intervene during earlier health care visits for children at risk for severe or fatal injury. Because head injuries account for over 80% of all suspected non-accidental injuries and over 90% of fatalities in the pediatric population, this intervention specifically targets all children ages 0-2 years who present in the Phoenix Children's Hospital (PCH) ED with a diagnosed head injury of any kind not resulting from a motor vehicle collision (MVC). These injuries include, but ae not limited to, abrasions, contusions, hematoma, ischemia, fractures, swelling or bruising. In this way, SunBrite expands the scope of detection for NAT to include injuries resulting from supervisory neglect.

PCH will implement the SunBrite pilot protocol in collaboration with key community partners who will be extensively involved in project design, implementation, and evaluation. In preparation for study recruitment, PCH and its partners will formalize the SunBrite process, create a curriculum, draft training tools to support the fidelity of SunBrite, finalize study materials (e.g., worksheets, data collection forms, interview scripts, consent documentation, and logic model), and conduct professional training. Once development is complete, pediatric patient families will be enrolled into the pilot program.

SunBrite study will utilize a simple, randomized, prospective study design, with 221 eligible pilot study participants randomized upon triage to one of two study arms: the control arm (73 families) or the treatment arm (148 families). Families in the control group will receive treatment as usual (TAU), which includes reporting to child welfare agencies when appropriate. In the treatment group, the patient/family will receive the SunBrite protocol, whose components include a screening, a brief intervention based in motivational interviewing (MI) techniques, and referral to treatment. All abuse and neglect, no matter the study arm, will be reported in accordance with hospital policy, federal and state laws.

All self-identified primary caregivers (legal guardians or parents) of children ages 0-2 who present in the PCH ED with a diagnosed intracranial injury will be automatically screened for eligibility. Caregivers will be initially screened by ED clinicians (e.g., physicians, nurse-practitioners) for eligibility based on age, injury (head), and method of injury (MOI) (non-MVC) using a standard clinical interview currently in place. All caregivers who screen positive based on these three criteria will then be deemed eligible for SunBrite. A trauma social worker will be notified by the ED that they have an eligible patient for consult. The social worker will meet the family and briefly describe the study and their eligibility. If they are willing to participate, the social worker will then obtain informed consent. All patient families will be fully consented in person in English or Spanish.

The screening, brief intervention, and referral to treatment will occur in the ED in the form of an abbreviated social work consultation prior to discharge. A social worker will complete an assessment for supervisory and household risks and then complete an injury risk worksheet to be used in the brief intervention. The social worker will engage caregivers in a 20- to 30-minute motivational interview (i.e., social work consult) using parent-coaching techniques for medical settings(12). In-person coaching facilitates active practice of these skills, supports further development of desired behaviors, and promotes long-term, sustainable risk mitigation.

The referral-to-treatment component of SunBrite identifies risks that may require further professional intervention, such as a history of trauma, mental illness, or substance abuse. For risks that warrant longer-term treatment, social workers will make referrals to external agencies and professionals for psychiatric evaluation, medication management, medically-assisted treatment (MAT), cognitive-behavioral therapy, and PTSD treatment.

Data from all participants, regardless of randomization, will be collected from patient health records. This will include patient demographics, injury characteristics, labs, imaging, consults, diagnoses, treatments, complications, and discharge notes. Patients will be followed for up to 12 months to assess study outcomes. The primary outcomes for this study are rates re-hospitalization (including frequency of hospitalization and length of stay) and return ED visits for any ICD-10 code. Secondary outcomes include complications from the indexed traumatic injury, other illnesses and conditions unrelated to trauma, and cost savings from reduced ED return visits and admissions. Based on PCH admissions data, we expect that 50% of eligible patients will return to the ED with an injury within one year of discharge. In addition to tracking all patients for 12 months post-discharge for any diagnosis at PCH, we will match our participants to the statewide database housed at the Arizona State University (ASU) Center for Health Information Research.

Quantitatively, we hypothesize that the proportion of patients measured on the primary outcome (return to ED) for the experimental group will be statistically smaller than the proportion in the control group under the following assumptions of a superiority design: 1) the percentage of patients that we expect to return to the ED is approximately 50% for the control group within one year of discharge to home and 25% for the experimental group; 2) the risk of type I error is alpha=.025; 3) power=.80. These parameters require a total sample size of 134 with a sample size of 67 for each group. However, we are planning to randomize in an unequal allocation of 2:1 to the experimental arm and oversample by 10%, bringing the total sample size up to 221 (148 in the experimental arm and 73 in the control arm). This design has an advantage in early phase trials, allowing investigators to explore treatment dimensions and optimize treatment utility.

We will also employ qualitative methods to provide rich feedback to enhance the implementation process and ensure project fidelity (e.g., identifying barriers and strategies to sustainability and wider dissemination). A formative evaluation of SunBrite will follow a plan, do, review, revise cycle of performance management that addresses the following intervention components: screening, staffing, brief intervention fidelity, referral, data collection, and reporting. . Quarterly advisory board meetings with community partners throughout the pilot program will provide an opportunity to update stakeholders on the pilot and receive feedback on implementation. Interviews with key stakeholders occurring at the start of the pilot, during program recruitment, and at the end of the recruitment process will provide important feedback to keep the pilot on track and achieve program goals. Voluntary interviews will assess experience with implementation and acceptability of SunBrite as implemented. Significantly, a research plan will be developed to validate SunBrite in a multi-site randomized trial.

To prepare for SunBrite information dissemination statewide, PCH will facilitate ongoing development of a formalized screening tool for use in EDs and manualize the SunBrite brief intervention and referral system. We will also design a dissemination plan (including funding) for SunBrite to incorporate a telemedicine option for the brief intervention. We will also disseminate findings from the pilot nationally through speaking engagements, conferences, posters, and published papers. In coordination with our community partners, we will develop a plan to sustain SunBrite in the PCH ED and to promote dissemination to other trauma centers.

ELIGIBILITY:
Inclusion Criteria

* Pediatric patients under the age of 2 presenting to the ED with intracranial trauma not resulting from a motor vehicle accident.
* Children admitted overnight for observation may be included in the study. Because of the age of the child, most children are held overnight or longer.

Exclusion Criteria

* Children with a head injury associated with a motor vehicle collision.
* Children whose guardian does not present in the ED with the patient at the time of admission.
* Children with developmental disabilities or autism.
* Medically fragile children, children with chronic illness, or children diagnosed with failure to thrive.
* Caregivers/guardians who do not speak English or Spanish

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2021-01 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Return visits to emergency department for any ICD-10 code | 12 months post enrollment
  Measured by the number of admissions to the ED as recorded in the patient's medical chart.

SECONDARY OUTCOMES:
Complications from traumatic head injury | 12 months post enrollment
  Any complications resulting from intracranial injury that child presents with in ED.
All illnesses and conditions of participant, including those unrelated to traumatic head injury | 12 months post enrollment
  Assessed via review of illnesses and conditions as recorded in the patient's medical chart.
Cost savings | 12 months post enrollment
  Savings resulting from reduced ED visits and readmissions to hospital.
Frequency of re-hospitalization | 12 months post enrollment
  Measured by number of hospital admissions as recorded in the patient's medical chart.
Hospital lengths of stay | 12 months post enrollment
  Measured in days as recorded in the patient's medical chart.

CONTACTS AND LOCATIONS:
Overall Officials: David M Notrica, MD, Principal Investigator — Phoenix Children's Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Louwers EC, Korfage IJ, Affourtit MJ, Scheewe DJ, van de Merwe MH, Vooijs-Moulaert FA, Woltering CM, Jongejan MH, Ruige M, Moll HA, De Koning HJ. Detection of child abuse in emergency departments: a multi-centre study. Arch Dis Child. 2011 May;96(5):422-5. doi: 10.1136/adc.2010.202358. Epub 2011 Jan 30. PMID 21278429
- [Result] King WK, Kiesel EL, Simon HK. Child abuse fatalities: are we missing opportunities for intervention? Pediatr Emerg Care. 2006 Apr;22(4):211-4. doi: 10.1097/01.pec.0000208180.94166.dd. PMID 16651907
- [Result] Bray JW, Del Boca FK, McRee BG, Hayashi SW, Babor TF. Screening, Brief Intervention and Referral to Treatment (SBIRT): rationale, program overview and cross-site evaluation. Addiction. 2017 Feb;112 Suppl 2:3-11. doi: 10.1111/add.13676. PMID 28074566